CLINICAL TRIAL: NCT07393594
Title: A Prospective, Multicenter, Observational Study Evaluating Serial T-ID Monitoring for the Prevention of CMV Disease and BK Virus-Associated Nephropathy Following Kidney Transplantation
Brief Title: Observational Study Evaluating Serial T-ID Monitoring -ID-ENTITY
Acronym: ID-ENTITY
Status: Not yet recruiting | Type: Observational
Sponsor: Transplant Genomics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: TGRP32 ID-ENTITY
Record Dates: First submitted 2026-01-30; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Kidney Diseases; Kidney Injury; BK Virus Infection; CMV; TTV Virus
Keywords: Biomarkers testing; Kidney transplant rejection; T-ID Assay; TRAC Assay cell free DNA; Biopsy
MeSH Terms: conditions — Kidney Diseases | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Blood tests, TRAC( cell free DNA) and T-ID — Blood collection

SUMMARY:
To evaluate the association between time-updated CMV and BK viral loads measured monthly by T-ID and the risk of CMV disease and/or biopsy-proven BK virus-associated nephropathy (BKVAN) during the first 12 months following kidney transplantation, accounting for the net immune environment (TTV viral load) and allograft injury (donor-derived cell-free DNA, dd-cfDNA).

DETAILED DESCRIPTION:
* To characterize time-updated viral detection patterns (e.g., transient vs sustained CMV or BK signals) identified by T-ID prior to development of CMV disease or BKVAN.
* To evaluate the clinical utility of T-ID monitoring, defined by the frequency and type of clinical management actions taken following test results.
* To estimate the diagnostic performance of T-ID for clinically meaningful viral infection compared with standard-of-care (PCR) testing and clinical adjudication.
* To quantify lead time between T-ID detection of viral cfDNA and standard-of-care confirmation or initiation of therapy.
* To assess the safety of biomarker-informed management, including both rejection following infection-directed management and infection following rejection-directed management.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet all the following criteria:

  * Written informed consent and HIPAA authorization obtained prior to any study-related data collection.
  * Age ≥18 years at the time of enrollment.
  * Recipient of a kidney transplant, including:
  * Primary or repeat kidney transplantation
  * Living-donor or deceased-donor transplantation
  * At 1 month post-kidney transplant at the time of enrollment.
  * Receiving maintenance immunosuppressive therapy per institutional standard of care.
  * Selected by the treating provider to undergo TRAC testing as part of usual post-transplant clinical monitoring.

Exclusion Criteria:

* Recipient of a combined organ transplant involving a non-renal solid organ (e.g., kidney-liver, kidney-heart) and/or islet cell transplantation.
* History of prior non-renal solid organ transplantation or islet cell transplantation.
* Known pregnancy at the time of enrollment.
* Known active viral infection at enrollment with any of the following:
* Hepatitis B surface antigen (HBsAg)-positive
* Hepatitis B virus (HBV) nucleic acid testing (NAT)-positive
* Human immunodeficiency virus (HIV) infection or HIV NAT-positive
* *Known active BK virus-associated nephropathy (BKVAN) or CMV disease at the time of enrollment.
* Medical, psychiatric, or social condition that, in the opinion of the Investigator, would interfere with the participant's ability to provide informed consent or comply with study procedures.
* Concurrent participation in another investigational biomarker study designed to evaluate clinical utility of post-transplant molecular diagnostics.

  * Participants with asymptomatic or low-level viral replication detected during routine clinical monitoring are eligible, provided there is no evidence of established CMV disease or BK virus-associated nephropathy at enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All subjects who meet eligibility criteria will be enrolled. As this is a non-interventional study, the protocol does not mandate any specific diagnostic, therapeutic, or management interventions. Clinical management decisions, including adjustments to immunosuppression, antiviral therapy, diagnostic testing, and biopsy decisions, remain entirely at the discretion of the treating clinicians.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2026-03-31 (Estimated); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-10-30 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint of the study is the time to first occurrence of either cytomegalovirus (CMV) disease or biopsy-proven BK virus-associated nephropathy (BKVAN) during the first 12 months post-kidney transplantation. | 12 Months
  * CMV disease will be defined according to standard clinical criteria, including CMV syndrome and/or tissue-invasive CMV disease, as determined by the treating clinician and documented in the medical record.
  * BK virus-associated nephropathy (BKVAN) will be defined as biopsy-proven BK virus nephropathy, characterized by histopathologic features consistent with BKVAN (including intranuclear viral inclusions and/or positive SV40 large T-antigen staining), in the setting of documented BK viral replication by standard-of-care testing (e.g., plasma or urine PCR).

IPD SHARING:
Plan to Share IPD: Undecided
All data collected will be analyzed and submitted to Journals publications.

REFERENCES:
- [Background] Clinical Utility of Peripheral Blood Gene Expression Profiling of Kidney Transplant Recipients to Assess the Need for Surveillance Biopsies in Subjects with Stable Renal Function January 2017 Journal of Transplantation Technologies & Research 07(03) DOI: 10.4172/2161-0991.1000177 Martin Roy First Thomas C Whisenant John Friedewald Show all 10 authors Michael M Abecassis Citations 6 Reads 239
- [Background] Arms MA, Fleming J, Sangani DB, Nadig SN, McGillicuddy JW, Taber DJ. Incidence and impact of adverse drug events contributing to hospital readmissions in kidney transplant recipients. Surgery. 2018 Feb;163(2):430-435. doi: 10.1016/j.surg.2017.09.027. Epub 2017 Nov 22. PMID 29174434
- [Background] Sinha R, Zhu Z, Park S, Rebello C, Kinsella B, Friedewald J, Kleiboeker S. Combined Metagenomic Viral Detection and Donor-Derived Cell-Free DNA Quantification in Plasma From Kidney Transplant Recipients. Transplant Proc. 2024 Jul-Aug;56(6):1522-1530. doi: 10.1016/j.transproceed.2024.06.003. Epub 2024 Jul 6. PMID 38972761
- [Background] Park S, Guo K, Heilman RL, Poggio ED, Taber DJ, Marsh CL, Kurian SM, Kleiboeker S, Weems J, Holman J, Zhao L, Sinha R, Brietigam S, Rebello C, Abecassis MM, Friedewald JJ. Combining Blood Gene Expression and Cellfree DNA to Diagnose Subclinical Rejection in Kidney Transplant Recipients. Clin J Am Soc Nephrol. 2021 Oct;16(10):1539-1551. doi: 10.2215/CJN.05530421. PMID 34620649
- [Background] Friedewald JJ, Kurian SM, Heilman RL, Whisenant TC, Poggio ED, Marsh C, Baliga P, Odim J, Brown MM, Ikle DN, Armstrong BD, Charette JI, Brietigam SS, Sustento-Reodica N, Zhao L, Kandpal M, Salomon DR, Abecassis MM, Clinical Trials in Organ T. Develop-ment and clinical validity of a novel blood-based molecular biomarker for subclinical acute rejection following kidney transplant. Am J Transplant. 2019;19(1):98-109. Epub 2018/07/10. doi: 10.1111/ajt.15011. PubMed PMID: 29985559; PMCID: PMC6387870
- [Background] Lo DJ, Kaplan B, Kirk AD. Biomarkers for kidney transplant rejection. Nat Rev Nephrol. 2014 Apr;10(4):215-25. doi: 10.1038/nrneph.2013.281. Epub 2014 Jan 21. PMID 24445740
- [Background] Bouamar R, Shuker N, Hesselink DA, Weimar W, Ekberg H, Kaplan B, Bernasconi C, van Gelder T. Tacrolimus predose concentrations do not predict the risk of acute rejection after renal transplantation: a pooled analysis from three randomized-controlled clinical trials(dagger). Am J Transplant. 2013 May;13(5):1253-61. doi: 10.1111/ajt.12191. Epub 2013 Mar 8. PMID 23480233
- [Result] Loupy A, Haas M, Roufosse C, Naesens M, Adam B, Afrouzian M, Akalin E, Alachkar N, Bagnasco S, Becker JU, Cornell LD, Clahsen-van Groningen MC, Demetris AJ, Dragun D, Duong van Huyen JP, Farris AB, Fogo AB, Gibson IW, Glotz D, Gueguen J, Kikic Z, Kozakowski N, Kraus E, Lefaucheur C, Liapis H, Mannon RB, Montgomery RA, Nankivell BJ, Nickeleit V, Nickerson P, Rabant M, Racusen L, Randhawa P, Robin B, Rosales IA, Sapir-Pichhadze R, Schinstock CA, Seron D, Singh HK, Smith RN, Stegall MD, Zeevi A, Solez K, Colvin RB, Mengel M. The Banff 2019 Kidney Meeting Report (I): Updates on and clarification of criteria for T cell- and antibody-mediated rejection. Am J Transplant. 2020 Sep;20(9):2318-2331. doi: 10.1111/ajt.15898. Epub 2020 May 28. PMID 32463180